CLINICAL TRIAL: NCT06037759
Title: Novel Cardiovascular Biomarkers in Patients With Kidney Disease
Acronym: CBKD
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: LHS0082
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Haemodialysis Complication; Major Adverse Cardiac Events
Keywords: Chronic Kidney Disease; End Stage Kidney Disease; Haemodialysis; Biomarkers; Major Adverse Cardiac Events
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Up to 30ml of blood will be collected for processing to serum or plasma/red cell pellet for downstream analysis.
  Novel Biomarkers: Galactin-3, cMyC, Troponin. Lipidomics Proteomics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases (N=50):: Patients with incident ESKD managed by HD (n=50)
  Interventions: Diagnostic Test: Cardiac Biomarkers; Diagnostic Test: Lipidomics; Diagnostic Test: Proteomics
- Controls (N=50): Patients with Incident ESKD managed by PD (n=20) Patients with CKD stage 3-4 (not on dialysis) with hypertension as a key risk factor for CKD and CVD (n=30)
  Interventions: Diagnostic Test: Cardiac Biomarkers; Diagnostic Test: Lipidomics; Diagnostic Test: Proteomics

INTERVENTIONS:
Diagnostic Test: Cardiac Biomarkers — Blood samples will be collected at baseline (within 6 weeks of dialysis start), at 6 months post-commencement and 12 months post-commencement of haemodialysis. The blood sampling will be mid-week samples taken at the dialysis start for haemodialysis patients, with a similar approach for the PD controls. For the CKD controls, the blood samples will be scheduled around routine clinic attendance, adhering where possible to the time intervals for HD cases and PD controls.
Diagnostic Test: Lipidomics — Blood samples will be collected at baseline (within 6 weeks of dialysis start), at 6 months post-commencement and 12 months post-commencement of haemodialysis. The blood sampling will be mid-week samples taken at the dialysis start for haemodialysis patients, with a similar approach for the PD controls. For the CKD controls, the blood samples will be scheduled around routine clinic attendance, adhering where possible to the time intervals for HD cases and PD controls.
Diagnostic Test: Proteomics — Blood samples will be collected at baseline (within 6 weeks of dialysis start), at 6 months post-commencement and 12 months post-commencement of haemodialysis. The blood sampling will be mid-week samples taken at the dialysis start for haemodialysis patients, with a similar approach for the PD controls. For the CKD controls, the blood samples will be scheduled around routine clinic attendance, adhering where possible to the time intervals for HD cases and PD controls.

SUMMARY:
Chronic kidney disease (CKD) is a long-term condition where the kidneys do not work as well as they should. End-stage kidney failure (ESKD) is the final, irreparable stage of chronic kidney disease (CKD), where kidney function has worsened, so the kidneys can no longer function independently.

At this stage, dialysis is required to remove waste products and excess fluid from the blood. There are two types of dialysis. In haemodialysis (HD), blood is pumped out of the body to an artificial kidney machine and returned to the body by tubes that connect a person to the machine. In peritoneal dialysis (PD), the inside lining of the belly acts as a natural filter. PD has the advantage of being gentler on the heart. HD causes significant stress to the heart by reducing the blood flow to the heart muscle, resulting in heart failure, irregular rhythms, and eventually sudden heart death. A large observational study showed that HD patients had 48% worse survival in the first two years than PD patients.

Several molecules ('biomarkers') can be detected in blood and inform doctors of heart damage. Studying the form and function of proteins (Proteomics), including how they work and interact with each other inside cells in patients, could help identify the onset of heart problems. HD patients are also prone to body fat changes (cholesterol/lipids). Due to high cholesterol, there is build-up on the walls of arteries, causing their hardening. In HD patients, this process is faster due to abnormalities in lipid structure. Therefore, studying the heart biomarkers, protein, and lipid makeup of HD patients may help to find people at substantial risk of heart and vascular problems and if they are likely to become unwell due to these heart problems.

DETAILED DESCRIPTION:
Currently, there is no specific approach to stratify CV risk in HD patients; therefore, patients are not offered targeted preventative interventions. This novel project will characterise circulating biomarkers and proteomics of myocyte damage, cardiac stress, fibrosis, and inflammation, including lipid composition. Understanding the cardiac biomarkers, targeted proteomics and lipidomics in HD patients as early predictors of CV outcomes will help better decisions on treatment choices and earlier interventions to improve outcomes in these patients. Proteomics and lipidomics, analysed with machine learning techniques, may offer new opportunities to improve risk stratification in these patients. The successful introduction of novel agents, comprising proprotein convertase subtilisin-like/kexin type 9 inhibitors, low-dose oral anticoagulants, sodium-glucose cotransporter 2 inhibitors, glucagon-like peptide-1 agonists, anti-inflammatory agents, and icosapent ethyl, offers an opportunity to reduce the burden of recurrent CV risk further based on their risk stratification. This study aims to obtain pilot data for promising cardiac biomarkers, proteomics and lipidomics, validating them against control groups and establishing prospective changes of the new markers and their relation to the major adverse cardiac events (MACE).

Study Objectives

1. To determine circulating plasma levels of new cardiac biomarkers (cMyC, galectin 3) in incident HD patients by comparing them to control groups (PD and CKD 3-4 (not on dialysis)) and to correlate with traditional biomarkers (hsTnT).
2. To evaluate the lipidome as a marker of CVD risk in incident HD patients by studying the indices of HDL quality and quantity, including HDL-particle number, HDL cholesterol, apolipoprotein (apo) A-I levels, serum amyloid A (SAA) content and HDL-cholesterol efflux capacity, and paraoxonase activity of apoB-depleted serum.
3. To evaluate proteomic signature as a marker of cardiac disease risk in incident HD patients by studying the proteomic platform of untargeted high-value proteins for CVD risk (as an exploratory analysis).
4. To explore the association between proposed cardiac biomarkers, proteomics, lipidome and MACE (as an exploratory analysis).

ELIGIBILITY:
Inclusion Criteria:

Patients aged≥45 years (or ≥18 with a history of diabetes). b. Cases: Incident haemodialysis patients c. A comparative arm of peritoneal dialysis patients and CKD 3-4 (not on dialysis) with hypertension as a key risk factor for CVD.

d. Capable of understanding the purpose and risks of the study, fully informed, and given informed consent.

Exclusion Criteria:

1. Patients with pre-existing heart disease will be excluded.
2. Patients with active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged ≥45 years (or ≥18 with a history of diabetes) for both cases and controls. Cardiovascular risk steeply increases after the age of 45 years. For this exploratory analysis, we intend to target patients at high risk of cardiovascular disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 12 months
  An exploratory analysis of all-cause mortality and Major Adverse Cardiac Events (MACE). MACE is defined as a composite of CV death, Ischemic Heart Disease (IHD), myocardial infarction (MI), stroke/TIA, Heart Failure, Cardiac revascularisation (percutaneous coronary intervention and coronary artery bypass graft), carotid endarterectomy. The follow-up will be 12 months for all patients. This will be correlated with biomarker, proteomic and lipidomic data.

CONTACTS AND LOCATIONS:
Overall Officials: Anirudh Rao, PhD, Principal Investigator — Liverpool University Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No
However, the samples will be bio-banked at Liverpool University Biobank which can be shared with researchers.